CLINICAL TRIAL: NCT00269295
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation, In-Patient Phase I/II Study to Determine the Safety and Immunogenicity of Ty800 in Healthy Adult Subjects
Brief Title: TY800 Dose Escalation (Typhoid)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-084
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-02

CONDITIONS: Typhoid and Paratyphoid Fevers
Keywords: Typhoid fever, S typhi, vaccine
MeSH Terms: conditions — Typhoid Fever; Paratyphoid Fever

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Cohort 1: Arm 1 (Experimental): 12 subjects to receive vaccine dose 1: 5 X 10^7 cfu.
  Interventions: Biological: Ty800
- Cohort 1: Arm 2 (Placebo Comparator): 6 subjects to receive placebo.
  Interventions: Drug: Placebo
- Cohort 2: Arm 1 (Experimental): 12 subjects to receive vaccine dose 2: 5 X 10^8 cfu.
  Interventions: Biological: Ty800
- Cohort 3: Arm 1 (Experimental): 12 subjects to receive vaccine dose 3: 5 X 10^9 cfu.
  Interventions: Biological: Ty800
- Cohort 3: Arm 2 (Placebo Comparator): 6 subjects to receive placebo.
  Interventions: Drug: Placebo
- Cohort 2: Arm 2 (Placebo Comparator): 6 subjects to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ty800 — Live attenuated Ty800 S typhi oral vaccine is co-administered with a sodium bicarbonate buffer solution. Dosages: 5 X 10^7 cfu, 5 X 10^8 cfu, and 5 X 10^9 cfu.
  Arms: Cohort 1: Arm 1; Cohort 2: Arm 1; Cohort 3: Arm 1
Drug: Placebo — 150 mL of the prepared sodium bicarbonate buffer solution. Placebo will look and taste essentially like the study product.
  Arms: Cohort 1: Arm 2; Cohort 2: Arm 2; Cohort 3: Arm 2

SUMMARY:
The purpose of this research study is to determine whether a new vaccine for typhoid fever is safe and effective. This study will also look at what effects (good and bad) this new vaccine, Ty800, has on the volunteers. The study will determine the highest dose of Ty800 that can be given without causing severe side effects. About 54 healthy males and females, ages 18-45 inclusive, in the Cincinnati metropolitan area will be enrolled in this study. They will be in the study for approximately 7 months, which includes a one month screening period, study product administration on Day 0, a 10-day hospital stay, an outpatient period on Days 9-28 with 4 follow-up visits, and safety follow-up phone calls at 2 and 6 months after hospital discharge. Researchers hope that this trial will help produce a vaccine that combines a high level of durable protective immunity with simplicity of administration and minimal reaction to the vaccine.

DETAILED DESCRIPTION:
Typhoid fever is a generalized infection of the reticuloendothelial system (spleen, liver, and bone marrow), gut-associated lymphoid tissue and gall bladder caused by Salmonella enterica serovar Typhi (S typhi). Humans are the only known natural host and reservoir for S typhi. Typhoid bacilli are transmitted by the fecal-oral route by contaminated drinking water or food. The ideal typhoid vaccine would combine high levels of durable protective immunity with simplicity of administration and minimal reactogenicity. The primary objective of this study is to assess the safety of Ty800 oral typhoid vaccine when administered as a single dose over a range of doses (5 x 10^7, 5 x 10^8, and 5 x 10^9 cfu) in healthy adult subjects compared to placebo. The primary endpoint is safety of Ty800 at the dose levels administered compared to placebo as determined by absence of bacteremia, absence of the diagnosis of typhoid fever as confirmed by a positive blood culture for the Ty800 vaccine organism, and by verifying that the null phoP/phoQ phenotype is retained by the isolated shed vaccine organism. Safety variables will be assessed by the reported incidence of adverse events (AE), blood cultures, and changes in vital signs, physical examination, and routine laboratory parameters over time at each vaccine dose level compared to placebo. The secondary objectives of this study are: to evaluate the immunogenicity of a single oral dose administration of Ty800 over a range of doses in healthy adult subjects; to evaluate the Ty800 vaccine dose response by comparing the immunogenicity profiles of each dose level; and to evaluate the shedding profile of Ty800 by determining the quantity and duration of shedding for each dose level. The tertiary objectives of this study include: evaluating, in a substudy, single nucleotide polymorphisms (SNPs) in candidate genes, e.g., IL-8 and interferon gamma, that may influence the immune response or persistent shedding of the vaccine organism and evaluating the induction of memory B cells in the vaccinated subjects. This study is a randomized, double-blind, placebo-controlled, dose escalation, inpatient phase I/II clinical trial. Three dose levels of Ty800 a vaccine will be evaluated and compared to placebo. Prior to randomization and administration of study vaccine, subjects will undergo screening evaluations. Healthy subjects meeting study eligibility criteria will be admitted to an inpatient facility with appropriate isolation containment the day prior to randomization, and they will remain in the unit for approximately 10 consecutive days. Three cohorts of 18 volunteers, representing 3 escalating doses of Ty800 typhoid vaccine will be challenged. In each cohort, 12 volunteers will receive Ty800 as a single oral dose, and 6 volunteers will receive placebo. Dose escalation will occur in a stepwise fashion and will be dependent upon the assessment of safety parameters and by meeting criteria for advancement to the next dose. Participants will be involved in study related procedures for up to 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women, aged 18 to 45 years, inclusive.
* Provide voluntary written informed consent prior to undergoing any study specific screening procedures.
* Must be willing to remain in the inpatient study unit for at least 10 days.
* Subjects must be of nonchildbearing potential, or if of childbearing potential (as determined by the investigator) must be using an effective licensed method of birth control (e.g., oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream, or foam; intrauterine contraceptive device; or Depo-Provera®; skin patch; vaginal ring or cervical cap or abstinence) for 30 days prior to vaccination and must agree to continue such precautions during the study and for 30 days after the final study visit. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., less than 1 percent per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner. ICH Guidance for Industry M3 Nonclinical Safety Studies for the Conduct of Human Clinical Trials for Pharmaceuticals (April 1997). If the subject uses abstinence as a method of birth control a questionnaire will be used to assure abstinence.
* Have normal screening laboratories for SGPT (ALT), creatinine, sodium, potassium, total white blood count (WBC), hemoglobin, neutrophils, lymphocytes, platelets, urine protein and hematuria.

Exclusion Criteria:

* Positive serum pregnancy test at screening or at admission (Day 1). Women who are pregnant or lactating and women of childbearing potential who do not agree to use acceptable birth control methods.
* History of immunocompromised states, human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome, autoimmune disease, leukemia, lymphoma, generalized malignancy, undergoing long-term chemotherapy, radiation therapy, or receiving systemic steroid therapy. A history of basal cell or squamous cell carcinoma cured by local excision more than 5 years ago will not be considered an exclusion criterion.
* Clinically significant history of cardiovascular disease, respiratory disease, gall bladder disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, sickle cell anemia, neurologic illness, psychiatric disorder requiring chronic medication or prior hospitalization.
* Presence of prosthetic cardiac valves or other intravascular or intra-articular prosthetic material.
* Presence of HIV antibody.
* Presence of hepatitis B surface antigen or hepatitis C antibody.
* HLA-B27 or IgA deficiency.
* Presence of Salmonella species and/or bacterial or parasitic pathogens in a screening stool examination.
* History of travel to a S typhi endemic area within the last 5 years, history of raising a child from a S typhi endemic area, vaccination against typhoid fever, infection with S typhi, or participation in a typhoid fever clinical trial using S typhi or an S typhi vector at any time. United States, Canada, Europe, New Zealand and Australia are not considered endemic areas.
* Clinically abnormal screening electrocardiogram (ECG) defined as pathologic Q waves and significant ST-T wave changes; criteria for left ventricular hypertrophy; and any nonsinus rhythm excluding isolated premature atrial contractions.
* Known allergy or sensitivity to 2 or more of the following antibiotics: ciprofloxacin, amoxicillin, trimethoprim-sulfamethoxazole, chloramphenicol, ceftriaxone, or quinolones (e.g., enoxacin, lomefloxacin, ofloxacin, norfloxacin).
* Known allergy to any components of the Ty800 vaccine or buffer (sodium bicarbonate/ascorbic acid).
* Receipt of blood/blood products or immunoglobulins within 6 months prior to the screening visit. Donation of blood within 2 months.
* A change in the subject's normal stool pattern within 3 months prior to screening visit. A normal stool pattern is defined as at least once a week and less than 4 times a day.
* Regular (monthly or more often) use of laxatives including herbal laxatives.
* Any medical illness requiring new prescription medication or hospitalization during the 45-day screening period prior to admission to the inpatient facility or have a temperature greater than or equal to 38.0ºC during the inpatient period prior to administering the study vaccine.
* Use of antibiotics within 7 days prior to study product administration.
* Use of any H2 receptor antagonists (e.g., Tagamet®, Zantac®, Pepcid®), proton pump inhibitors (e.g., Prilosec® OTC, Protonix®, and Prevacid®), or prescription acid suppression medication or over-the-counter (OTC) antacids within 72 hours of study product administration.
* Subjects who are commercial food handlers, day care workers, or health care workers involved in direct patient contact. Subjects with young children (<2 years) at home or with household contacts who are immunocompromised, pregnant, or breast-feeding.
* Participation in any other investigational drug, device, or vaccine trial within the 30 days prior to screening or planned participation within 30 days after the final study visit.
* Subjects who are unable to pass a written test that describes typhoid fever and explains the requirements of the clinical trial.
* Any other condition or responsibility, such as a medical, psychiatric, or social condition or occupational responsibility that, in the judgment of the investigator, would interfere with or serve as a contradiction to the subject's participation in the protocol or assessment of the investigational product.
* Subjects who smoke and cannot stop smoking for the duration of the inpatient study. -Subjects will be excluded if their screening laboratory test results fall outside of the laboratory normal range with the exception that 1) WBC and neutrophil counts below the laboratory normals will be allowable if they are in keeping with the levels seen in a condition that is prevalent in our population known as benign ethnic neutropenia, 2) transaminase levels (ALT) below the lower limit of "normal" will also not be an exclusion criterion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Assess the safety of Ty800 oral typhoid vaccine when administered as a single dose over a range of doses (5 x 10^7, 5 x 10^8, 5 x 10^9 cfu) in healthy adult subjects compared to placebo. | Duration of study.

SECONDARY OUTCOMES:
To evaluate the shedding profile of Ty800 by determining the quantity and duration of shedding for each dose level. Spread of the vaccine organism to placebo subjects will also be monitored as an outcome variable. | Days 1-8, 11, 14, and 28.
To evaluate the immunogenicity of the single oral dose administration of Ty800 over a range of doses in healthy adult subjects. | At intervals after vaccination between Days 7 through 28.
To evaluate the Ty800 vaccine dose response by comparing the immunogenicity profiles of each dose level. | At intervals after vaccination between Days 7 through 28.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States